CLINICAL TRIAL: NCT00537693
Title: Cytokine Removal by CRRT in Pediatric Sepsis: A Comparison of Convection Versus Diffusion
Brief Title: Cytokine Removal by CRRT in Pediatric Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Dialysis Solutions Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-21133
Record Dates: First submitted 2007-09-27; First posted 2007-10-01 (Estimated); Last update posted 2010-09-02 (Estimated); Status verified 2010-09

CONDITIONS: Sepsis
Keywords: Continuous Renal Replacement Therapy (CRRT); Sepsis; Convection; Diffusion
MeSH Terms: conditions — Sepsis | interventions — Continuous Renal Replacement Therapy

ARMS (2):
- 1 (Active Comparator): CRRT via Convection
  Interventions: Procedure: Continuous Renal Replacement Therapy
- 2 (Active Comparator): CRRT via Diffusion
  Interventions: Procedure: Continuous Renal Replacement Therapy

INTERVENTIONS:
Procedure: Continuous Renal Replacement Therapy — Patients will be randomized to either arm for the first 24 hours of the study and then crossover to the second arm for the second 24 hours of the study.

SUMMARY:
This pilot study will compare the effect of diffusive versus convective Continuous Renal Replacement Therapy (CRRT) in children with sepsis who require CRRT.

The hypothesis for the study is that convective forms of CRRT provide enhanced clearance of cytokines and improved clinical responses as compared to a diffusive CRRT modality.

DETAILED DESCRIPTION:
The purpose of this study is to test the hypothesis that convective forms of Continuous Renal Replacement Therapy (CRRT) provides enhanced clearance of cytokines compared to a diffusive CRRT modality. Also, we plan to test the hypothesis that patients who receive convective CRRT modalities demonstrate improved clinical responses to patients who receive a diffusive CRRT modality.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented sepsis or suspected SIRS
* Patients initiating CRRT
* Age 1 to 21 years

Exclusion Criteria:

* Patients on ECMO
* Patients receiving concomitant plasma exchange
* Cardiopulmonary bypass procedure within 96 hours of CRRT
* Patients with new onset acute leukemia
* Patients with active autoimmune disease
* Ungrafted stem cell transplant recipients

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
A 25% additional decrease in IL-6 concentration change | The First 24 hours of CRRT

SECONDARY OUTCOMES:
Other cytokine removal rates | First 24 hours of CRRT
Cytokine absorption on the CRRT membrane | First 24 hours of CRRT
Hemodynamic parameters | First 24 hours of CRRT
Changes in serum cytokine concentrations and clearance | After crossover, from 24-48 hours
Changes in serum cytokine concentrations | From beginning to end of the study, independent of modality

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Goldstein, MD, Principal Investigator — Baylor College of Medicine
Locations (5):
- United States (5):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Helen De Vos Children's Hospital, Grand Rapids, Michigan
  - Texas Childrens Hospital, Houston, Texas